CLINICAL TRIAL: NCT01726699
Title: Scripps Tumorgraft Study
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Applied Genetic Epidemiology, Scripps Translational Science Institute
Other Study IDs: 12-6011
Record Dates: First submitted 2012-11-06; First posted 2012-11-15 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Solid Tumor Malignancy or Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer Diagnosis

SUMMARY:
Study the genetic traits of cancerous tissues and to help improve cancer treatment by developing tumor models for studying new cancer drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or over
* diagnosis of a solid tumor malignancy, either resectable or metastatic or a hematologic malignancy
* cognitively and emotionally able to give informed consent

Exclusion Criteria:

* Under age 21
* Not cognitively or emotionally able to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a solid tumor malignancy or a hematologic malignancy
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Facilitate the development of individualized tumorgraft models for many different types of cancer. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura Goetz, MD, Principal Investigator — Director, Applied Genetic Epidemiology
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States